CLINICAL TRIAL: NCT03136016
Title: Design of a School Randomized Trial for Nudging Students Towards Healthy Diet and Physical Activity
Brief Title: Nudging, Healthy Diet and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, Full professor, Rio de Janeiro State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: nudgingpaappas
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (No Intervention): without any activity
- educational activities (Experimental): The students will receive educational activities in the classroom.
  Interventions: Behavioral: educational activities
- nudging (Experimental): The students will receive changes in the school environment (nudge strategies);
  Interventions: Behavioral: nudging
- nudging + educational activities (Experimental): The students will receive educational activities and changes in the school environment.
  Interventions: Behavioral: nudging + educational activities

INTERVENTIONS:
Behavioral: educational activities — Group 2 will receive classroom-based educational activities based on an earlier study, called PAPPAS, which was developed in the same city and constituted a school-based intervention with the objective of reducing the consumption of sweetened beverages and biscuits and increase the consumption of fruits, vegetables and beans
  Arms: educational activities
Behavioral: nudging — In group 3, changes in the environment will be included that will facilitate both physical activity and healthy food choices
  Arms: nudging
Behavioral: nudging + educational activities — Group 4 will receive both interventions
  Arms: nudging + educational activities

SUMMARY:
The present study is a randomized school-based trial of a sample of 5th and 6th grade students from 10 public schools in the municipality of Duque de Caxias, metropolitan area of Rio de Janeiro, Brazil. The aim is to investigate whether adding nudging actions to the intervention group of PAAPPAS trial (PAAPAS Study, NCT02711488) increase fruits, vegetables and water consumption and daily energy expenditure, in a factorial design.

ELIGIBILITY:
Inclusion Criteria:

5th and 6th grades students consent form signed by parents/tutors

Exclusion Criteria:

pregnant girls

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 6 months
  Sample size of PAAPPAS Nudge was calculated based on a minimum effect of 0.15 in BMI variation and considering intra and intergroup comparisons. Body mass index (BMI) will be determined as a ratio between body weight (kg) and squared height (m).

SECONDARY OUTCOMES:
Fruit consumption | 6 months
  Food intake will be assessed by a food frequency questionnaire validated for teenagers in Rio de Janeiro and one 24-hour recall (Rec24h). Netbooks containing a computer program developed for school use, based on a technique called "Multiple Pass Method" will be used.
Vegetable consumption | 6 months
  Vegetable consumption will be assessed by one 24-hour recall (Rec24h). The food items in the Rec24h will be transformed into daily consumption and grouped according to similary in nutritional containing
Water consumption | 6 months
  Water consumption will be assessed by a question regarding the number of glasses of water consumed during a day. Glasses of water consumed during a day will be assessed by a question at baseline and at the end of the study.
Physical activity | 6 months
  Physical activity levels will be measured through a validated questionnaire including six questions about frequency and time of different physical activities domains.

CONTACTS AND LOCATIONS:
Locations (1):
- 10 Schools of Metropolitan Area, Duque de Caxias, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antunes ABS, Hassan BK, Pinto RL, Sichieri R, Cunha DB. A choice architecture intervention targeting school meals and water frequency intake: A school-based randomized trial. Appetite. 2024 Feb 1;193:107118. doi: 10.1016/j.appet.2023.107118. Epub 2023 Nov 17. PMID 37977257